CLINICAL TRIAL: NCT01911832
Title: Impact of Widths After Gastric Tube Reconstruction on Quality of Life for Patients With Esophagogastric Cancers
Brief Title: Impact of Gastric Tube Reconstruction Widths on Quality of Life for Esophagogastric Cancers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Professor of the West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WqLE-201324
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
Keywords: Cancer of the esophagogastric junction; Reconstruction of gastric tube; Quality of life; Width; Regurgitation
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gastrectomy and subtotal gastrectomy (Experimental): to compare the quality of life between esophagojejunostomy after total gastrectomy(TG group) and Roux-en-Y gastrojejunostomy after subtotal gastrectomy(SG group)
  Interventions: Procedure: esophagojejunostomy after total gastrectomy; Procedure: Roux-en-Y gastrojejunostomy after subtotal gastrectomy
- Wide and narrow reconstruction tube (Experimental): to compare the quality of life between wide tube reconstruction after subtotal gastrectomy(WG group) and narrow tube reconstruction after subtotal gastrectomy(NG group) in Roux-en-Y gastrojejunostomy
  Interventions: Procedure: wide tube reconstruction after subtotal gastrectomy; Procedure: narrow tube reconstruction after subtotal gastrectomy

INTERVENTIONS:
Procedure: esophagojejunostomy after total gastrectomy
  Other Names: total gastrostomy group(TG group)
  Arms: Gastrectomy and subtotal gastrectomy
Procedure: Roux-en-Y gastrojejunostomy after subtotal gastrectomy
  Other Names: subtotal gastrectomy(SG group)
  Arms: Gastrectomy and subtotal gastrectomy
Procedure: wide tube reconstruction after subtotal gastrectomy
  Other Names: wide gastric tube group(WG group)
  Arms: Wide and narrow reconstruction tube
Procedure: narrow tube reconstruction after subtotal gastrectomy
  Other Names: narrow gastric tube group(NG group)
  Arms: Wide and narrow reconstruction tube

SUMMARY:
The incidence of cancer of the esophagogastric junction has rapidly risen in recent three decades, and surgery still remains the optimum therapy. For Siewert's type II and III cancer, esophagojejunostomy after total gastrectomy and Roux-en-Y gastrojejunostomy after subtotal gastrectomy are regarded as the two main surgical approaches. Esophagojejunostomy after total gastrectomy brings high survival rate and low local recurrence rate which may also induces pulmonary infection or regurgitation. Roux-en-Y gastrojejunostomy after subtotal gastrectomy needs reconstruction of the gastric tube and the width of reconstruction tube was a key factor to predicate prognosis. However, no evidence supplies a comprehensive standard on the width of reconstruction tube which often ranges from 3 cm to 6 cm. Both narrow and wide reconstruction tubes have their own advantages and disadvantages. So the prospective trail recruits patients into three groups: total gastrostomy group (TG group), wide gastric tube group (WG group) and narrow gastric tube group (NG group). And the investigators compare the quality of life using integrated questionnaire of QLQ-STO22 and QLQ-C30 and related symptom relief as main endpoints.

DETAILED DESCRIPTION:
With the decreasing prevalence of gastric cancer, the incidence of cancer of the esophagogastric junction has rapidly risen in recent three decades, especially in North America and Europe. Despite the use of chemotherapy, its 5-year survival rate is still low (less than 30%) for cancer of the esophagogastric junction. Surgery still remains the optimum therapy for cancer of the esophagogastric junction. For Siewert's type II and III cancer, esophagojejunostomy after total gastrectomy and Roux-en-Y gastrojejunostomy after subtotal gastrectomy are regarded as the two main surgical approaches. For quality of life, no prospective trial provides evidence comparing the two approaches.

With a complete clearance of lymph nodes, esophagojejunostomy after total gastrectomy brings high 5-year survival rate, and can decrease the rate of local recurrence. However, due to the whole gastrectomy, the patients often represent bile regurgitation which may induce pulmonary infection, regurgitation asthma and weight loss.

Roux-en-Y gastrojejunostomy after subtotal gastrectomy reserve partial gastric body which was reconstructed into gastric tube. The remaining gastric body still peristalses and functions as well as a stomach. At the same time, the remaining gastric body keeps acid-secreting function which may induce acid regurgitation after surgery.

For Roux-en-Y gastrojejunostomy after subtotal gastrectomy, the width of reconstruction gastric tube was a key factor to predicate prognosis, and it often ranges from 3 cm to 6 cm, without universal standard. Narrow gastric tube may lack enough blood supply, as a result, it increase the rate of anastomotic leakage. On the contrary, wide gastric tube takes up much thoracic capacity which may disturb the normal pulmonary and cardiovascular function. Tabira and his colleagues conduct a prospective trail that proves the width of gastric tube has no relevance to local blood supply, anastomotic leakage and postoperative nutrition, but the study lack enough patients which may increase bias. So, there is no reliable evidence to predict the quality of postoperative life.

The prospective trail recruits patients with of cancer of the esophagogastric junction. And eligible patients were assigned into three groups: total gastrostomy group (TG group), wide gastric tube group (WG group) and narrow gastric tube group (NG group). Quality of life include integrated questionnaire of QLQ-STO22 and QLQ-C30 and related symptom relief was assessed as primary endpoint. And local recurrence, disease free survival, metastatic rate, overall survival and short-term complication of surgery were also observed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed esophagogastric cancers
2. age between 18 to 80 years
3. no evidence of metastasis of adjacent organs
4. organs function well to tolerate surgery
5. no special treatment before surgery
6. informed consent was written

Exclusion Criteria:

1. with other site tumor,simultaneously
2. locally recurrent gastric or esophageal cancer
3. had a history of malignant tumor within 5 years(except the skin cancer)
4. pregnant or lactating women
5. there was contraindication for operation
6. discovery of metastasis in the operation
7. with mental disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
quality of life | 3 years
  quality of life include: 1)integrated questionnaire of QLQ-STO22 and QLQ-C30. 2)related symptom relief of regurgitation, dysphagia and heartburn et al.

SECONDARY OUTCOMES:
local recurrence | 1 year
disease free survival | 1 year
  the time from operation to confirmed local recurrence, distant metastases, or death due to disease or treatment, whichever occurred first
metastatic rate | 1 year
  ratio of the patients with metastasis after the operation
overall survival | 1 and 3 years
  the fraction of the person from the operation the death,no matter the reason of the death.
short-term complication of the surgery | first 30 day after operation
  complication including pulmonary infection, bleeding and anastomotic leakage et al.

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Background] Vial M, Grande L, Pera M. Epidemiology of adenocarcinoma of the esophagus, gastric cardia, and upper gastric third. Recent Results Cancer Res. 2010;182:1-17. doi: 10.1007/978-3-540-70579-6_1. PMID 20676867
- [Background] Hasegawa S, Yoshikawa T. Adenocarcinoma of the esophagogastric junction: incidence, characteristics, and treatment strategies. Gastric Cancer. 2010 Jun;13(2):63-73. doi: 10.1007/s10120-010-0555-2. Epub 2010 Jul 3. PMID 20602191
- [Background] Allum WH, Stenning SP, Bancewicz J, Clark PI, Langley RE. Long-term results of a randomized trial of surgery with or without preoperative chemotherapy in esophageal cancer. J Clin Oncol. 2009 Oct 20;27(30):5062-7. doi: 10.1200/JCO.2009.22.2083. Epub 2009 Sep 21. PMID 19770374
- [Background] Mariette C, Piessen G, Briez N, Gronnier C, Triboulet JP. Oesophagogastric junction adenocarcinoma: which therapeutic approach? Lancet Oncol. 2011 Mar;12(3):296-305. doi: 10.1016/S1470-2045(10)70125-X. Epub 2010 Nov 23. PMID 21109491
- [Background] Johansson J, Djerf P, Oberg S, Zilling T, von Holstein CS, Johnsson F, Walther B. Two different surgical approaches in the treatment of adenocarcinoma at the gastroesophageal junction. World J Surg. 2008 Jun;32(6):1013-20. doi: 10.1007/s00268-008-9470-7. PMID 18299921
- [Background] Ielpo B, Pernaute AS, Elia S, Buonomo OC, Valladares LD, Aguirre EP, Petrella G, Garcia AT. Impact of number and site of lymph node invasion on survival of adenocarcinoma of esophagogastric junction. Interact Cardiovasc Thorac Surg. 2010 May;10(5):704-8. doi: 10.1510/icvts.2009.222778. Epub 2010 Feb 13. PMID 20154347
- [Background] De Giacomo T, Francioni F, Venuta F, Trentino P, Moretti M, Rendina EA, Coloni GF. Complete mechanical cervical anastomosis using a narrow gastric tube after esophagectomy for cancer. Eur J Cardiothorac Surg. 2004 Nov;26(5):881-4. doi: 10.1016/j.ejcts.2004.07.024. PMID 15519175
- [Background] Matsuda T, Kaneda K, Takamatsu M, Takahashi M, Aishin K, Awazu M, Okamoto A, Kawaguchi K. Reliable preparation of the gastric tube for cervical esophagogastrostomy after esophagectomy for esophageal cancer. Am J Surg. 2010 May;199(5):e61-4. doi: 10.1016/j.amjsurg.2009.08.046. Epub 2010 Mar 3. PMID 20202621
- [Background] Pierie JP, de Graaf PW, van Vroonhoven TJ, Obertop H. The vascularization of a gastric tube as a substitute for the esophagus is affected by its diameter. Dis Esophagus. 1998 Oct;11(4):231-5. doi: 10.1093/dote/11.4.231. PMID 10071804
- [Background] Tabira Y, Sakaguchi T, Kuhara H, Teshima K, Tanaka M, Kawasuji M. The width of a gastric tube has no impact on outcome after esophagectomy. Am J Surg. 2004 Mar;187(3):417-21. doi: 10.1016/j.amjsurg.2003.12.008. PMID 15006575